CLINICAL TRIAL: NCT02429895
Title: A Phase 2, Multicenter, Open-Label Extension (OLE) Study With ABT-122 in Active Psoriatic Arthritis Subjects Who Have Completed a Preceding Study M14-197 Phase 2 Randomized Controlled Trial (RCT)
Brief Title: A Phase 2, Multicenter Open-Label Extension (OLE) Study With ABT-122 in Active Psoriatic Arthritis Subjects Who Have Completed a Preceding Study M14-197
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal business decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-198; 2014-005527-27 (EudraCT Number)
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Psoriatic Arthritis
Keywords: Methotrexate; Efficacy; Safety
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — ABT-122

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (open-label extension) (Experimental): All subjects will start treatment with ABT-122
  Interventions: Drug: ABT-122

INTERVENTIONS:
Drug: ABT-122 — Injection

SUMMARY:
A Phase 2, Multicenter, Open-Label Extension (OLE) Study with ABT-122 in Active Psoriatic Arthritis Subjects Who Have Completed a Preceding Study M14-197 Phase 2 Randomized Controlled Trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed preceding Study M14-197 (ABT-122) RCT study and have not developed any discontinuation criteria of Study M14-197.
2. If female, subject must meet one of the following criteria:

   * Postmenopausal (defined as no menses for at least 1 year).
   * Surgically sterile (bilateral oophorectomy or hysterectomy)

   If subject does not meet one of the above two categories, subject must use one of the following methods of birth control, from the time of the first dose of study drug until 150 days after the last dose of study drug:
   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation started at least 2 months prior to the first dose of study drug: oral, intravaginal or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation started at least two months prior to randomization: oral, injectable, or implantable
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion/ligation
   * Be with a vasectomized partner (procedure at least 6 months earlier, the vasectomized male partner should be your sole partner)
   * Sexual abstinence (refraining from heterosexual intercourse during the entire study period)
3. If male, subject must be surgically sterile (have had a vasectomy more than 6 months prior to Screening) or must be practicing at least 1 of the following methods of birth control from the time of the first dose of study drug until 150 days post last dose of study drug:

   * Subject using condom and female partner(s) using an intrauterine device (IUD);
   * Subject using condom and female partner(s) using hormonal contraceptives (oral, vaginal, parenteral or transdermal);
   * Subject using condom and female partner(s) using double-barrier method (contraceptive sponge; diaphragm or vaginal ring with spermicidal jellies, creams, or spermicide);
   * Total abstinence from sexual intercourse as the preferred lifestyle of the subject; periodic abstinence is not acceptable.
   * Subject must also agree to not donate sperm starting on the first day of study drug administration until 150 days after the last dose of study drug.
4. Subjects must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any study-specific procedures.
5. Subject is judged to be in good health as determined by the Investigator.

Exclusion Criteria:

1. Pregnant or breastfeeding or plans to become pregnant during study participation.
2. Ongoing infections at Day 1 (Week 0) that have NOT been successfully treated within 14 days.
3. Anticipated requirement or receipt of any live vaccine during study participation including up to 120 days after the last dose of study drug.
4. Current enrollment in another investigational study; with the exception of Study M14-197, which is required.
5. Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to continue to receive ABT-122.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR) 20 response rate by visit | From Week 0 to Week 24
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
American College of Rheumatology (ACR) 50 response rate by visit | From Week 0 to Week 24
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
American College of Rheumatology (ACR) 70 response rate by visit | From Week 0 to Week 24
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
Change in American College of Rheumatology (ACR) the individual component by visit | From Week 0 to Week 24
  ACR criteria measure improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant.
Change in Disease Activity Score DAS28 [hsCRP] by visit | From Week 0 to Week 24
  Determine by disease activity score using 28 joint counts (DAS28) and high-sensitivity C-reactive protein (hsCRP) lab test.
Change in Psoriatic Disease Activity Score (PASDAS) by visit | From Week 0 to Week 24
  PASDAS determined by tender or swollen joint counts, patient reported outcome and hsCRP lab test.
Change in Psoriasis Area and Severity Index (PASI) by visit | From Week 0 to Week 24
  Determined by scores for the amount and severity of a patient's psoriasis.
Change in Psoriasis Target Lesion Score by visit | From Week 0 to Week 24
  Determined by plaque erythema, plaque scaling and plaque thickness scores.
Change in Dactylitis Assessment by visit | From Week 0 to Week 24
  Determined by presence of dactylitis, swelling, and tenderness in each digit of both hands and both feet.
Change in Enthesitis Sites Comprising the Total Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index by visit | From Week 0 to Week 24
  Determined by the presence and severity of enthesitis.
Change in Self-Assessment of Psoriasis Symptoms (SAPS) by visit | From Week 0 to Week 24
  Determined by scores given by patients regarding the severity of their psoriatic symptoms.
Change in skin biopsy/biomarkers | From Week 0 to Week 24
  Optional samples to assess changes related on disease activity/prognosis of psoriatic arthritis (PsA), autoimmunity/inflammation, and/or response to anti-PsA medications.
Change in the quality of life, function and work as measured by the Short-Form Health Survey Version 2.0 (SF36v2) by visit | From Week 0 to Week 24
  Quality of life are self reported measures to assess the physical function of the patient and how their activities are impacted by their disease.
Change in the quality of life, function and work as measured by Bath AS Disease Activity Index (BASDAI) by visit | From Week 0 to Week 24
  Quality of life are self reported measures to assess the physical function of the patient and how their activities are impacted by their disease.
Change in the quality of life, function and work as measured by the Fatigue Numeric Rating Scale by visit | From Week 0 to Week 24
  Quality of life are self reported measures to assess the physical function of the patient and how their activities are impacted by their disease.
Change in the quality of life, function and work as measured by the Sleep Quality Scale by visit | From Week 0 to Week 24
  Quality of life are self reported measures to assess the physical function of the patient and how their activities are impacted by their disease.

CONTACTS AND LOCATIONS:
Overall Officials: Heikki T Mansikka, MD, Study Director — AbbVie
Locations (36):
- Site Reference ID/Investigator# 138922, Woolloongabba, Australia
- Bulgaria (6):
  - Site Reference ID/Investigator# 138925, Plovdiv
  - Site Reference ID/Investigator# 138926, Plovdiv
  - Site Reference ID/Investigator# 138927, Plovdiv
  - Site Reference ID/Investigator# 138928, Sofia
  - Site Reference ID/Investigator# 138930, Sofia
  - Site Reference ID/Investigator# 138929, Sofia
- Czechia (3):
  - Site Reference ID/Investigator# 138934, Prague
  - Site Reference ID/Investigator# 138933, Prague
  - Site Reference ID/Investigator# 138932, Uherské Hradiště
- Germany (2):
  - Site Reference ID/Investigator# 141365, Frankfurt
  - Site Reference ID/Investigator# 138953, Lübeck
- Site Reference ID/Investigator# 138959, Budapest, Hungary
- Latvia (4):
  - Site Reference ID/Investigator# 138983, Ādaži
  - Site Reference ID/Investigator# 138985, Riga
  - Site Reference ID/Investigator# 138982, Riga
  - Site Reference ID/Investigator# 138984, Valmiera
- New Zealand (3):
  - Site Reference ID/Investigator# 138986, Auckland
  - Site Reference ID/Investigator# 138988, Nelson
  - Site Reference ID/Investigator# 138987, Newtown, Wellington
- Poland (12):
  - Site Reference ID/Investigator# 139000, Bialystok
  - Site Reference ID/Investigator# 139012, Bydgoszcz
  - Site Reference ID/Investigator# 138999, Elblag
  - Site Reference ID/Investigator# 139007, Katowice
  - Site Reference ID/Investigator# 139006, Krakow
  - Site Reference ID/Investigator# 139005, Lublin
  - Site Reference ID/Investigator# 139026, Oświęcim
  - Site Reference ID/Investigator# 139004, Poznan
  - Site Reference ID/Investigator# 139001, Stalowa Wola
  - Site Reference ID/Investigator# 139011, Szczecin
  - Site Reference ID/Investigator# 139003, Torun
  - Site Reference ID/Investigator# 139010, Wroclaw
- Romania (2):
  - Site Reference ID/Investigator# 139013, Bucharest
  - Site Reference ID/Investigator# 139016, Targu-Mures, Jud. Mures
- Spain (2):
  - Site Reference ID/Investigator# 139022, Elche
  - Site Reference ID/Investigator# 139020, Santiago de Compostela

REFERENCES:
- [Derived] Genovese MC, Weinblatt ME, Mease PJ, Aelion JA, Peloso PM, Chen K, Li Y, Liu J, Othman AA, Khatri A, Mansikka HT, Leszczynski P. Dual inhibition of tumour necrosis factor and interleukin-17A with ABT-122: open-label long-term extension studies in rheumatoid arthritis or psoriatic arthritis. Rheumatology (Oxford). 2018 Nov 1;57(11):1972-1981. doi: 10.1093/rheumatology/key173. PMID 30032191